CLINICAL TRIAL: NCT05627037
Title: Evaluation of the Marginal Bone Level of Titanium Implants Produced by Additive Manufacture, in 30 and 90 Days: Randomized Within-subject Clinical Trial of 1-year Non-inferiority
Brief Title: Marginal Bone Level Around Titanium Implants Produced by Additive Manufacture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Plenum (M3 Health Industria e Comercio de Produtos Médicos) (Unknown)
Responsible Party: Principal Investigator, Giuseppe Alexandre Romito, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 59844422.4.0000.0075
Record Dates: First submitted 2022-10-31; First posted 2022-11-25 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Dental Implants
Keywords: implant, osseointegration
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: Split-Mouth Study Model
Who Masked: Care Provider, Outcomes Assessor
Masking Description: either the operator or the patient will be blinded for the primary outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loading in 30 days (Experimental): Implant allocated to the study arm will be restored with a temporary restoration after 30 days of implant placement, that will be replaced with definitive restoration after 90 days of implant placement.
  Interventions: Device: Dental implant produced by additive manufacture
- Loading in 90 days (Active Comparator): Implant allocated to the study arm will be restored directly with the definitive restoration after 90 days of implant placement.
  Interventions: Device: Dental implant produced by additive manufacture

INTERVENTIONS:
Device: Dental implant produced by additive manufacture — In a split-mouth setup, each participant will receive two implants in the posterior region of the mandible or maxilla. After implant insertion, one implant will be randomly allocated to receive Temporary restoration after 30 days and definitive restoration after 90 days
  Arms: Loading in 30 days
Device: Dental implant produced by additive manufacture — In a split-mouth setup, each participant will receive two implants in the posterior region of the mandible or maxilla. After implant insertion, one implant will receive definitive restoration after 90 days
  Arms: Loading in 90 days

SUMMARY:
The aim of this study will be to evaluate the non-inferiority of implants produced by additive manufacture loaded in 30 days when compared with those loaded in 90 days, in relation to marginal bone loss, after 01 (one) year of follow-up

DETAILED DESCRIPTION:
This randomized Split-mouth clinical study of non-inferiority will monitor for one year partially edentulous patients in the posterior region of the mandible or maxilla, rehabilitated with 2 implants (AM) in the same Arch to evaluate the success rate of the implant, one loaded at 30 days after installation and the other at 90 days. Changes in marginal bone level and osseointegration success will be evaluated, with visits and data collection in 0 days (baseline), 30 days, 90 days, 6 months and 1 year

ELIGIBILITY:
Inclusion Criteria:

* Patients treated and referred by the Dental Clinic of the School of Dentistry of the University of São Paulo;
* Individuals over 18 years and under 70 years of age;
* Good general health;
* signed Informed Consent Form;
* Need for rehabilitation with dental implants in areas of mandible or posterior maxilla (premolars and/or molars);
* bacterial plaque index ≤ 20% (Silness & Loe, 1964);
* bleeding rate of ≤ 20% (Loe & Silness, 1963);
* Sufficient alveolar bone volume for an implant of:

  * Length: 8 or 10mm
  * Diameter: 3.5mm, 4. 00mm or 4. 5mm
* Bone quality type I-III;
* No associated bone regeneration.

Exclusion Criteria:

* Pregnant and lactating women;
* Uncontrolled diabetes;
* History of chemotherapy or radiotherapy in the last 5 years;
* Radiotherapy in areas of the head and neck;
* Use of immunosuppressants, bisphosphonate or prolonged use of corticosteroids;
* Smokers;
* Alcohol or drug abuse;
* Untreated periodontitis;
* History of previous bone increase in the implant installation region;
* Presence of residual roots at the site receiving the implant;
* Bone density type IV
* Individuals with connective tissue disorders or metabolic diseases;
* Postmenopausal osteoporosis or other systemic diseases that may affect bone metabolism;
* Need for guided bone regeneration at the time of implant installation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Loss (MBL) | 1 year
  Digital periapical radiographs will be taken at the implant installation (baseline) after 1 year. The radiographs will be taken using the parallelism technique with a positioner that supports the digital sensor in order to standardize the radiographs.

SECONDARY OUTCOMES:
Implant success rate | 1 year
  The success rate or failure of each implant in clinical and radiographic findings will be classified using the success criteria defined by Buser et al. (1990)
  1. Absence of persistent subjective complaints, such as pain, foreign body sensation and/or dysesthesia.
  2. Absence of a recurrent peri-implant infection with suppuration.
  3. Absence of mobility.
  4. Absence of a continuous radiolucency around the implant.
  5. Possibility for restoration. These criteria will be monitored at 0 days (baseline), 30 days, 90 days, 6 months, and the final endpoint is one year
Modified Plaque Index (mPI) | 1 year
  Modified Plaque Index (Mombelli, Van Oosten Et.Al 1987):
  Scoring Criteria:
  Score 0: No detection of plaque Score 1:Plaque only recognized by running a probe across the smooth marginal surface of the implant Score 2: Plaque can be seen by the naked eye. Score 3: Abundance of soft matter. The changes in Modified Plaque Index (mPI) will be monitored at 0 days (baseline), 30 days, 90 days, 6 months, and the final endpoint is one year
Modified Bleeding Index (mBI) | 1 year
  Modified Sulcus Bleeding Index (Mombelli, Van Oosten Et.Al 1987):
  Scoring Criteria:
  Score 0: No bleeding when probe is passed along the gingival margin. Score 1: Isolated bleeding, spots present. Score 2: Blood forms a confluent red line on margins. Score 3: Heavy or profuse bleeding. The changes in Modified Bleeding Index (mBI) will be monitored by a blinded calibrated examiner at 0 days (baseline), 30 days, 90 days, 6 months, and the final endpoint is one year
Pocket probing depth (PPD) | 1 year
  Pocket Probing Depth (PPD) will be measured by a blinded calibrated Examiner, and The changes in Pocket Probing Depth (PPD) will be monitored at 0 days (baseline), 30 days, 90 days, 6 months, and the final endpoint is one year
clinical attachment level (CAL) | 1 year
  Clinical attachment level (CAL) will be measured by a blinded calibrated Examiner, and The changes in clinical attachment level (CAL) will be monitored at 0 days (baseline), 30 days, 90 days, 6 months, and the final endpoint is one year

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe A Romito, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Dentistry - University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No